CLINICAL TRIAL: NCT05485285
Title: Peculiarities of Pain in Patients With Mine-explosive Wounds Depending on the Localization of the Wound at the Stages of Treatment
Acronym: PPPM-EWDL
Status: Completed | Type: Observational
Sponsor: Bogomolets National Medical University (Other)
Responsible Party: Principal Investigator, Vasyl' Horoshko, Chief researcher, Bogomolets National Medical University
Other Study IDs: №158 (23.05.2022)
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Chronic Pain
Keywords: pain, wounds, stages of treatment
MeSH Terms: conditions — Chronic Pain; Pain; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- retrospective analysis: A retrospective analysis of disease histories for the period from 2014 to 2021 was carried out. Data collection was carried out at all stages of treatment: medical and nursing brigade, military mobile hospital, military medical clinical center, during rehabilitation, within 12 months of the injury.
  Interventions: Other: visual analog scale
- prospective study: Recruitment of patients for the prospective study was carried out in the period from 02.24.2022 to 05.24.2022
  Interventions: Other: visual analog scale

INTERVENTIONS:
Other: visual analog scale — Data collection was carried out at all stages of treatment: medical and nursing brigade, military mobile hospital, military medical clinical center, during rehabilitation, within 12 months of the injury.
  Other Names: neuropathic pain Didier Bouhassiraa (DN4).; Chaban Quality of Life Scale; The Hospital Anxiety and Depression Scale (HADS); Mississippi PTSD scale (military version)

SUMMARY:
Mine-explosive wounds in the general structure of combat sanitary losses reach 25%. They are characterized by significant damage resulting in high intensity pain. In patients who received mine-explosive injuries in the conditions of hostilities, such pain has its own unique features. It is necessary to pay more attention to the problem of pain treatment in patients of this category, because about 87.2% of cases have negative results of treatment - it becomes chronic.

DETAILED DESCRIPTION:
Over the last ten years, the amount of pathology caused by mine-explosive devices has increased significantly. Mine-explosive wounds in the general structure of combat sanitary losses reach 25%. They often have a combined character. Such an injury must be considered as a multifactorial injury resulting from the combined impact on a person of a shock wave, gas jets, flames, toxic products, fragments of the hull, secondary projectiles, which cause severe injuries in the area of direct damage and the body as a whole. Mine-explosive injuries are characterized by multiple, combined or combined injuries with a high degree of severity - 8-10%. Also, even in peacetime, terrorists often use powerful explosive devices. Here, the mortality rate is 10-20% of the total number of injured, and 80-90% suffer from the consequences - mine-explosive injuries. Compared to the wars of the past, the number of seriously wounded with combined injuries has increased to 25-30%. This is primarily due to the use of high-precision ammunition and mine-explosive ammunition. In general, multiple and combined damage in local conflicts today is 25-62%. Lethality in case of mine-explosive injury reaches 37-41.4%. The mortality rate among the wounded with mine-explosive injuries who were admitted to the stage of qualified medical care was 17.4%, more than half of the wounded died as a result of blood loss. In 63.7%, death occurs in the first 24 hours after injury.The direct and most frequent causes are shock and blood loss (49.1%), destruction of vital organs (28.4%). About 90% of all combat deaths occur before the wounded reaches the first stage of treatment.

The peculiarities of pain in patients with mine-explosive wounds depending on the localization of the wound at the stages of treatment need to be studied, because the subjective feelings and emotional experiences experienced by patients during the wounding in combat conditions through the prism of psychological disorders have their own characteristics. Since in 87.2% of cases it is not possible to achieve a positive result of treatment, the data of our study will play an important role in their treatment.

ELIGIBILITY:
Inclusion Criteria:

* the presence of gunshot wounds

Exclusion Criteria:

* no gunshot wounds

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients were injured during hostilities
Sampling Method: Probability Sample
Enrollment: 660 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
visual analog scale | 12 months
  from 0 to 10 points
Didier Bouhassiraa DN4 | 12 months
  4 or more points (a neuropathic pain component is present)
The Hospital Anxiety and Depression Scale | 12 months
  0-7 is the norm 8-13 - mild depressive disorders 14-18 - depressive disorders of medium severity 19-22 - severe depressive disorders 23 and more - depressive disorders of a very severe degree of severity
Chaban Quality of Life Scale | 12 months
  up to 56 inclusive - a very low level 57-66 - low 67-75 - average 76-82 - tall 83-100 is very high
Mississippi PTSD scale (military version) | 12 months
  the mean values of the total score are 76±18 for well-adjusted servicemen, 86±26 for servicemen with mental disorders, and 130±18 for those with PTSD

CONTACTS AND LOCATIONS:
Locations (1):
- Bogomolets National Medical University, Ministry of Health of Ukraine, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided
I plan to share